CLINICAL TRIAL: NCT04822714
Title: Sequential Exploratory Mixed Method in Developing and Evaluating the Effectiveness of Mobile-phone Career Competencies Intervention for Malaysian Public Sector Managers
Brief Title: Effectiveness of Mobile-phone Career Competencies Intervention for Malaysian Public Sector Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Public Service Department Malaysia (Unknown)
Responsible Party: Principal Investigator, Ho Hsin Hung, Principal Investigator/ Senior Assistant Secretary, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPM
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Competency-Based Education; Competence
Keywords: career competencies; mobile career intervention; career behavioral action

STUDY DESIGN:
Intervention Model Description: This study is a single blind, multiple center parallel, randomized control trial (RCT) design incorporate individual treatment to all the participants with the mobile career competencies intervention aim to enhance the career competencies among the participants
Who Masked: Participant
Masking Description: The participants was blinded during the recruitment and allocation via electronic consent format and the intervention conducted through mobile intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Career Competencies Intervention (Experimental): The intervention protocol has five main components and is designed in English language. The first component consists of an educational session. The second component focuses on one's reflection on motivation and qualities. The third component assists users in working out strategies with others. The fourth component prompts users to reflect on and narrate their emerging career stories through goal-setting identification activities. The fifth component includes the government's human resource practices, training programs offered, and policies. The fourth and fifth component require users to reflect on their work exploration and career control career competencies.
  Interventions: Behavioral: Mobile Career Competencies Intervention
- Waitlist control (No Intervention): Waitlist control group attended work and basic training from the organization as usual. They only receive the mobile intervention after the intervention group completing of the intervention.

INTERVENTIONS:
Behavioral: Mobile Career Competencies Intervention — Mobile career competencies intervention aim to enhance the career competencies (career behavioral action) among the participants
  Arms: Mobile Career Competencies Intervention

SUMMARY:
This study aims to evaluate the effectiveness of a user and expert centric mobile phone-based career intervention program of career competencies among Malaysian public managers.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a user and expert centric mobile phone-based career intervention program of career competencies among Malaysian public managers. In this study, the Social Cognitive Career Theory (SCCT) is adopted as the framework to develop mobile phone-based intervention for career competencies. There is two phases in the study whereby in Phase 1, a qualitative approach developing the components in the career intervention module and mobile phone application features. Phase 2 that evaluates the mobile phone-based career intervention program. Validation will be conducted to meet the objectives of (i) the usability of the mobile communication career intervention application (survey), and (ii) evaluation of the effectiveness of the intervention program for career competencies delivered through mobile phone application (randomized controlled trial). The primary outcome of this study is career competencies. The career competencies score will be compared between participants in the intervention and control group at the baseline, and follow-ups at week four and week 12 respectively, using mixed design ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Must be Administrative and Diplomatic Officers (ADO) who use mobile application (Android)
* Must be in Grade 41
* Informed consent obtained

Exclusion Criteria:

* The officer that use IPhone
* The officer that involved in disciplinary issues

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Career Competencies | 12 weeks
  assessed by Career Competencies Questionnaire - 1=low career competencies & 5=high career competencies
Validation of Mobile Career Competencies Intervention | 1 week
  Assessed by USE Questionnaire - 1 Very Not Useful & 5 Very Useful
  * Usefulness
  * Ease of Use
  * Ease of Learning
  * System Satisfaction

SECONDARY OUTCOMES:
Reflection on motivation | 12 weeks
  subscale of career competencies and assessed by Career Competencies Questionnaire - 1=low reflection on motivation & 5=high reflection on motivation
Reflection on qualities | 12 weeks
  subscale of career competencies and assessed by Career Competencies Questionnaire - 1=low reflection on qualities& 5=high reflection on qualities
Networking | 12 weeks
  subscale of career competencies and assessed by Career Competencies Questionnaire - 1=low networking & 5=high networking
Self-profiling | 12 weeks
  subscale of career competencies and assessed by Career Competencies Questionnaire - 1=low self-profiling & 5=high self-profiling
Work exploration | 12 weeks
  subscale of career competencies and assessed by Career Competencies Questionnaire - 1=low work exploration & 5=high work exploration
Career control | 12 weeks
  subscale of career competencies and assessed by Career Competencies Questionnaire - 1=low career control & 5=high career control

CONTACTS AND LOCATIONS:
Overall Officials: Hsin Hung Ho, Master, Principal Investigator — Public Service Department Malaysia
Locations (1):
- Public Service Department Malaysia, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsin Hung, H., & Roziah, M. R. (2019). A Systematic Literature Review on the Competencies fo Public Services. International Conference on Educational Research and Practice 2019 (ICERP 2019), UPM, 57.
- [Background] Ho, H. H., Foo, C. N., & Baki, R. (2019). Training but no Training. International Journal of Academic Research in Business & Social Sciences, 9(7), 77-87.
- [Result] Ho HH, Mohd Rasdi R, Ibrahim R, Md Khambari MN. Developing and evaluating the effectiveness of mobile phone-based career intervention for career competencies of Malaysian public managers: Protocol for a mixed method study. Internet Interv. 2020 Sep 3;22:100349. doi: 10.1016/j.invent.2020.100349. eCollection 2020 Dec. PMID 32995304